CLINICAL TRIAL: NCT04371081
Title: Amplatzer Piccolo Occluder Japan Post-marketing Database Surveillance
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Japanese society of Congenital Interventional Cardiology (Unknown)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10290
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Amplatzer Piccolo Occluder: Amplatzer Piccolo Occluder device implant
  Interventions: Device: Amplatzer Piccolo Occluder

INTERVENTIONS:
Device: Amplatzer Piccolo Occluder — Interventional placement of vascular occluder

SUMMARY:
The purpose of this post-marketing clinical use database surveillance is to observe the frequency, type, and degree of adverse device effects and adverse events in order to assure the safety of the medical device, and to collect safety and efficacy information for evaluating the results of its clinical use.

DETAILED DESCRIPTION:
The Surveillance will be conducted per the standards required by the Ministry of Health, Labour and Welfare (MHLW) and in the standards for post-marketing surveillances and studies [except for those defined in the Ministerial Ordinance on Good Clinical Practice for Medical Devices (MHLW Ordinance No. 36, 2005)] based on Paragraph 4, Article 23-2-9 (including application mutatis mutandis per Article 23-2-19 of Revised PAL) of the Law on Securing Quality, Efficacy and Safety of Pharmaceuticals and Medical Devices, etc. (Law No. 145, 1960, hereinafter referred to as "Revised PAL") by the Marketing Authorization Holder or accredited foreign manufacturer of a medical device defined in Paragraph 1, Article 23-2-5 of Revised PAL.

ELIGIBILITY:
Inclusion Criteria:

The device is used to percutaneously close the PDA of a patient who meets all of the following:

* PDA ≤4 mm in diameter
* PDA ≥3 mm in length
* Weight ≥700 g

Exclusion Criteria:

* Age <3 days
* Coarctation of the aorta
* Left pulmonary artery stenosis
* Cardiac output that is dependent on right to left shunt through the PDA due to pulmonary hypertension
* Thrombus in the implant site, or sign of venous thrombus in a vessel in which the occluder is inserted and delivered
* Endocarditis, or infection that can cause bacteremia
* Allergic or potentially allergic to nickel

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with patent ductus arteriosus (PDA) in whom an Amplatzer™ Piccolo Occluder (Piccolo) implant was attempted will be included in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The rate of major complications through 180 days after an attempted Piccolo device implant | Through 180 days after an attempted Piccolo device implant
The rate of effective closure of the ductus arteriosus among subjects with a successful Piccolo implant as assessed by the presence of either a Grade 0 or Grade 1 shunt at the 6-month follow-up by transthoracic echocardiography | At the 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Showa University Hospital, Tokyo, Japan